CLINICAL TRIAL: NCT04865198
Title: Role of Neuralized1 and RGS14 Genes With ASD Patients
Brief Title: Neuralized1 and RGS14 Genes
Status: Completed | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Yusuf Ozkul, Professor, TC Erciyes University
Other Study IDs: NEURL1RGS14
Record Dates: First submitted 2021-04-20; First posted 2021-04-29 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Autism Spectrum Disorder; High-functioning Autism; Healthy
Keywords: ASD; High Functioning Autism; NEURL1; RGS14; Gene expression
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — In this study, 2 ml of peripheral blood was taken from each subject. RNA was isolated from peripheral blood followed by cDNA synthesis. RNA and cDNA samples of the subjects were preserved.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with Autism Spectrum Disorder (ASD): Patients diagnosed with ASD in a child psychiatry clinic.
  Interventions: Diagnostic Test: Neurl1 gene expression; Diagnostic Test: RGS14 gene expression
- Patients with High Functioning Autism (HFA): Patients diagnosed with ASD in a child psychiatry clinic and with an IQ above 70.
  Interventions: Diagnostic Test: Neurl1 gene expression; Diagnostic Test: RGS14 gene expression
- Healty control: Healthy volunteers who are in the age range compatible with the patient groups.
  Interventions: Diagnostic Test: Neurl1 gene expression; Diagnostic Test: RGS14 gene expression

INTERVENTIONS:
Diagnostic Test: Neurl1 gene expression — This observational case control study. The gene expression was examined.
Diagnostic Test: RGS14 gene expression — This observational case control study. The gene expression was examined.

SUMMARY:
Autism is a broad spectrum neurodevelopmental disease. Some individuals with ADS by high cognitive functions are diagnosed with High Functioning Autism (HFA). In some studies, it has been shown that NEURL1 gene increases learning and memory and RGS14 gene is suppressed them. We aimed to evaluate the differences between the expression levels of these genes between ASD, HFA and healthy controls and the role of these genes in the pathogenesis of ASD. Patients with 20 ASD and 20 HFA, and 20 healthy controls compatible with patient ages were included in this study. Expression of NEURL-1 and RGS14 genes was evaluated by quantitative Real Time PCR (qRT-PCR).

DETAILED DESCRIPTION:
ASD is a neurological disease starting in the early stages of life and is characterized by cognitive and behavioral disorders (Ansel et al., 2008;Alvares et al., 2020). It is considered that the etiology of ASD stems from genetic, epigenetic and environmental factors; however, it has not yet been definitively clarified(Ito et al., 2017).

we aimed to evaluate the differences between the expression levels of these genes between ASD, HFA and healthy controls and the role of these genes in the pathogenesis of ASD.

Method:

Patients with ASD (n=20) and HFA (n=20), and healthy controls (n=20) compatible with patient ages were included in this study. Clinical evaluations of the patients were made and classification was made in accordance with DSM-IV diagnostic criteria.

High Pure RNA Isolation Kit (Roche Diagnostic, Version 12, Germany) was used for RNA isolation. cDNA synthesis was performed from these RNAs with the ranscriptor High Fidelity cDNA Synthesis Kit (Roche Diagnostics, GmbH, Mannheim).

qRT-PCR was performed using the LightCycler®480 Real Time Ready Assay Master Probe Kit (Roche Diagnostics, GmbH, Mannheim).The incubation was made with the PCR device program for 10 minutes at 95oC for 45 cycles, for 10 sec at 95oC, and for 60 sec at 60oC. The Ct values were obtained from the Light Cycler 480 Software Program, and both genes were analyzed separately. The comparative CT method (2-ΔΔCT) was used to determine the relative quantification of target genes, normalized to a housekeeping gene (β-actin).

Statisticaly:

The results of the experiments were evaluated using R 3.1.1 (www.r-project.org). and Chi-Square Tests, Mann-Whitney U-Test, Kruskal-Wallis H-Tests. The P<0.05 level was taken as significant.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed ASD or HFA patient,
* Being between the ages of 2-16.

Exclusion Criteria:

* To use medicine,
* Have a other syndromic illness,
* Being younger than 2 years old or over 16 years old.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Group 1: Patients diagnosed with ASD in a child psychiatry clinic. Group 2: Patients diagnosed with HFA in a child psychiatry clinic. Group 3: Healty controls
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-01-10 (Actual); Primary Completion 2014-08-30 (Actual); Study Completion 2014-08-30 (Actual)

PRIMARY OUTCOMES:
NEURL1 gene expression levels | Two months
  After RNA isolation from blood samples of the subjects, NEURL1 gene expression was studied by QPCR method. The 2-ΔΔCT method was applied for the relative quantification of the samples that were normalized with ACTB.
RGS14 gene expression levels | Two months
  After RNA isolation from blood samples of the subjects, RGS14 gene expression was studied by QPCR method. The 2-ΔΔCT method was applied for the relative quantification of the samples that were normalized with ACTB.

SECONDARY OUTCOMES:
Age | an average of 1 year
  Age of subjects
Gender | an average of 1 year
  Gender (male/female) of subjects
Intellectual disability (ID) | an average of 1 year
  Intellectual disability is when a person has certain limitations in cognitive functioning and skills, including communication, social and self-care skills.It was determined according to DSM-IV diagnostic criteria and clinical evaluation.
Consanguinity | an average of 1 year
  Relationships of consanguinity between subjects were evaluated in terms of pathogenesis of the disease.
Presence of Neurological Disease in Relatives | an average of 1 year
  In the presence of a neurological disease in relatives, its relationship with the pathogenesis of the disease was evaluated.
Corelation tests | an average of 1 year"
  The relationships of the clinical and demographical findings in the study groups with the genes were evaluated statistically.

CONTACTS AND LOCATIONS:
Overall Officials: Hamiyet Eciroğlu, Phd. St., Principal Investigator — Alanya Alaaddin Keykubat University; Elif F. Şener, Assoc. Prof., Principal Investigator — TC Erciyes University; Didem B. Öztop, Assoc. Prof., Principal Investigator — Ankara University; Sevgi Özmen, Assoc. Prof., Principal Investigator — TC Erciyes University; Dilek Kaan, Phd., Principal Investigator — TC Erciyes University; Yusuf Özkul, Prof. Dr., Study Chair — TC Erciyes University

IPD SHARING:
Plan to Share IPD: Undecided
The details and reports of the study will be shared after the article is published.

REFERENCES:
- [Background] Ansel A, Rosenzweig JP, Zisman PD, Melamed M, Gesundheit B. Variation in Gene Expression in Autism Spectrum Disorders: An Extensive Review of Transcriptomic Studies. Front Neurosci. 2017 Jan 5;10:601. doi: 10.3389/fnins.2016.00601. eCollection 2016. PMID 28105001
- [Background] Charman T, Baird G. Practitioner review: Diagnosis of autism spectrum disorder in 2- and 3-year-old children. J Child Psychol Psychiatry. 2002 Mar;43(3):289-305. doi: 10.1111/1469-7610.00022. PMID 11944873
- [Background] Ito H, Morishita R, Nagata KI. Autism spectrum disorder-associated genes and the development of dentate granule cells. Med Mol Morphol. 2017 Sep;50(3):123-129. doi: 10.1007/s00795-017-0161-z. Epub 2017 May 22. PMID 28534217
- [Background] Rao PA, Beidel DC, Murray MJ. Social skills interventions for children with Asperger's syndrome or high-functioning autism: a review and recommendations. J Autism Dev Disord. 2008 Feb;38(2):353-61. doi: 10.1007/s10803-007-0402-4. Epub 2007 Jul 20. PMID 17641962
- [Background] Sener EF, Cikili Uytun M, Korkmaz Bayramov K, Zararsiz G, Oztop DB, Canatan H, Ozkul Y. The roles of CC2D1A and HTR1A gene expressions in autism spectrum disorders. Metab Brain Dis. 2016 Jun;31(3):613-9. doi: 10.1007/s11011-016-9795-0. Epub 2016 Jan 19. PMID 26782176
- [Background] Misra V. The social brain network and autism. Ann Neurosci. 2014 Apr;21(2):69-73. doi: 10.5214/ans.0972.7531.210208. PMID 25206065
- [Background] Sullivan JM, De Rubeis S, Schaefer A. Convergence of spectrums: neuronal gene network states in autism spectrum disorder. Curr Opin Neurobiol. 2019 Dec;59:102-111. doi: 10.1016/j.conb.2019.04.011. Epub 2019 Jun 18. PMID 31220745
- [Background] O'Brien G, Pearson J. Autism and learning disability. Autism. 2004 Jun;8(2):125-40. doi: 10.1177/1362361304042718. PMID 15165430
- [Background] Landsiedel J, Williams DM, Abbot-Smith K. A Meta-Analysis and Critical Review of Prospective Memory in Autism Spectrum Disorder. J Autism Dev Disord. 2017 Mar;47(3):646-666. doi: 10.1007/s10803-016-2987-y. PMID 28116668
- [Background] Vellano CP, Lee SE, Dudek SM, Hepler JR. RGS14 at the interface of hippocampal signaling and synaptic plasticity. Trends Pharmacol Sci. 2011 Nov;32(11):666-74. doi: 10.1016/j.tips.2011.07.005. Epub 2011 Sep 8. PMID 21906825
- [Background] Lamsa K, Lau P. Long-term plasticity of hippocampal interneurons during in vivo memory processes. Curr Opin Neurobiol. 2019 Feb;54:20-27. doi: 10.1016/j.conb.2018.08.006. Epub 2018 Sep 5. PMID 30195105
- [Background] Zeithamova D, Schlichting ML, Preston AR. The hippocampus and inferential reasoning: building memories to navigate future decisions. Front Hum Neurosci. 2012 Mar 26;6:70. doi: 10.3389/fnhum.2012.00070. eCollection 2012. PMID 22470333
- [Background] Besag FM. Epilepsy in patients with autism: links, risks and treatment challenges. Neuropsychiatr Dis Treat. 2017 Dec 18;14:1-10. doi: 10.2147/NDT.S120509. eCollection 2018. PMID 29296085
- [Background] Richter JD. Cytoplasmic polyadenylation in development and beyond. Microbiol Mol Biol Rev. 1999 Jun;63(2):446-56. doi: 10.1128/MMBR.63.2.446-456.1999. PMID 10357857
- [Result] Jacobs D, Steyaert J, Dierickx K, Hens K. Physician View and Experience of the Diagnosis of Autism Spectrum Disorder in Young Children. Front Psychiatry. 2019 May 28;10:372. doi: 10.3389/fpsyt.2019.00372. eCollection 2019. PMID 31191373
- [Result] Goh S, Peterson BS. Imaging evidence for disturbances in multiple learning and memory systems in persons with autism spectrum disorders. Dev Med Child Neurol. 2012 Mar;54(3):208-13. doi: 10.1111/j.1469-8749.2011.04153.x. Epub 2012 Jan 23. PMID 22269006
- [Result] Pavlopoulos E, Trifilieff P, Chevaleyre V, Fioriti L, Zairis S, Pagano A, Malleret G, Kandel ER. Neuralized1 activates CPEB3: a function for nonproteolytic ubiquitin in synaptic plasticity and memory storage. Cell. 2011 Dec 9;147(6):1369-83. doi: 10.1016/j.cell.2011.09.056. PMID 22153079
- [Result] Jaagura M, Taal K, Koppel I, Tuvikene J, Timmusk T, Tamme R. Rat NEURL1 3'UTR is alternatively spliced and targets mRNA to dendrites. Neurosci Lett. 2016 Dec 2;635:71-76. doi: 10.1016/j.neulet.2016.10.041. Epub 2016 Oct 22. PMID 27780737
- [Result] Taal K, Tuvikene J, Rullinkov G, Piirsoo M, Sepp M, Neuman T, Tamme R, Timmusk T. Neuralized family member NEURL1 is a ubiquitin ligase for the cGMP-specific phosphodiesterase 9A. Sci Rep. 2019 May 8;9(1):7104. doi: 10.1038/s41598-019-43069-x. PMID 31068605
- [Result] Lee SE, Simons SB, Heldt SA, Zhao M, Schroeder JP, Vellano CP, Cowan DP, Ramineni S, Yates CK, Feng Y, Smith Y, Sweatt JD, Weinshenker D, Ressler KJ, Dudek SM, Hepler JR. RGS14 is a natural suppressor of both synaptic plasticity in CA2 neurons and hippocampal-based learning and memory. Proc Natl Acad Sci U S A. 2010 Sep 28;107(39):16994-8. doi: 10.1073/pnas.1005362107. Epub 2010 Sep 13. PMID 20837545
- [Result] Squires KE, Gerber KJ, Pare JF, Branch MR, Smith Y, Hepler JR. Regulator of G protein signaling 14 (RGS14) is expressed pre- and postsynaptically in neurons of hippocampus, basal ganglia, and amygdala of monkey and human brain. Brain Struct Funct. 2018 Jan;223(1):233-253. doi: 10.1007/s00429-017-1487-y. Epub 2017 Aug 3. PMID 28776200
- [Result] Martin KC, Casadio A, Zhu H, Yaping E, Rose JC, Chen M, Bailey CH, Kandel ER. Synapse-specific, long-term facilitation of aplysia sensory to motor synapses: a function for local protein synthesis in memory storage. Cell. 1997 Dec 26;91(7):927-38. doi: 10.1016/s0092-8674(00)80484-5. PMID 9428516
- [Result] Hosoda N, Funakoshi Y, Hirasawa M, Yamagishi R, Asano Y, Miyagawa R, Ogami K, Tsujimoto M, Hoshino S. Anti-proliferative protein Tob negatively regulates CPEB3 target by recruiting Caf1 deadenylase. EMBO J. 2011 Apr 6;30(7):1311-23. doi: 10.1038/emboj.2011.37. Epub 2011 Feb 18. PMID 21336257
- [Result] Evans PR, Parra-Bueno P, Smirnov MS, Lustberg DJ, Dudek SM, Hepler JR, Yasuda R. RGS14 Restricts Plasticity in Hippocampal CA2 by Limiting Postsynaptic Calcium Signaling. eNeuro. 2018 Jun 4;5(3):ENEURO.0353-17.2018. doi: 10.1523/ENEURO.0353-17.2018. eCollection 2018 May-Jun. PMID 29911178
- See also: American Psychiatric Association. Diagnostic and statistical manual of mental disorders — https://books.google.com.tr/books?id=-JivBAAAQBAJ&printsec=frontcover&redir_esc=y#v=onepage&q&f=false